CLINICAL TRIAL: NCT02024997
Title: Improving Pancreas Radiotherapy Plans Using Respiration-driven Anatomic Deformation: A Pilot Study
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Wensha Yang, PhD., Assistant Professor, Cedars-Sinai Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: IIT2012-07-YANG-MRIRESP
Record Dates: First submitted 2013-12-18; First posted 2013-12-31 (Estimated); Last update posted 2014-10-30 (Estimated); Status verified 2014-10

CONDITIONS: Pancreatic Cancer
Keywords: Pancreatic malignancy; Radiation Therapy
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Abdominal MRI (Experimental): Subjects will undergo magnetic resonance imaging (MRI) with contrast. Magnetic resonance (MR)_freebreathing scan will be acquired. MR_inspiration scan will be acquired. MR_expiration scan will be acquired.
  Interventions: Other: Magnetic Resonance Imaging (MRI)

INTERVENTIONS:
Other: Magnetic Resonance Imaging (MRI)

SUMMARY:
The overall aim of this study is to investigate a novel "dual instance" planning method to make use of the respiratory motion to improve pancreatic radiation therapy (RT) treatment planning.

Specific Aim 1: Acquire patient abdominal MRI and CT at both deep inspiration (INSP) and expiration (EXP) positions and characterize the changes in geometric relationships between the INSP and EXP instances for tumor and normal tissues including stomach, duodenum and bowel. We hypothesize that INSP and EXP MRI and CT characterization will allow identification of patients who may benefit from the dual instance planning method.

Specific Aim 2: Develop, investigate and evaluate plans based on free breathing, single instance breath hold, and the novel dual instance anatomical information. We hypothesize that use of the dual instance method will lead to improved plans, demonstrated by the ability to increase dose to the target, while maintaining the clinically-accepted normal tissue dose constraints.

ELIGIBILITY:
Inclusion Criteria:

* Any patient with a biopsy proven diagnosis of malignancy involving the pancreas to be treated with radiation therapy
* Age >18 years
* Ability to understand and the willingness to sign a written informed consent document
* Creatinine or creatinine clearance of <1.5 times the upper limit of normal or >45 mL/min/1.73m2 for patients with creatinine levels above normal. Modification of Diet in Renal Disease (MDRD) formula was used to calculate the creatinine level

Exclusion Criteria:

* Patients who are currently receiving any investigational agents
* Unable to undergo MRIs
* Patients with late stage kidney disease or who have had a liver transplant
* Individuals who are allergic to animal dander or have asthma that may be enflamed by proximity to animals will be excluded as the scans will take place in a facility where animal research is also performed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2013-01; Primary Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Compare magnetic resonance (MR) in different breath-hold phases to quantify respiration induced anatomic changes | Baseline only (at least 3 days after CT simulation and up to 1 week after the initiation of radiation treatment)

SECONDARY OUTCOMES:
Modeling the feasibility of the dose escalation using respiration induced anatomic changes | Baseline only (at least 3 days after CT simulation and up to 1 week after the initiation of radiation treatment)

CONTACTS AND LOCATIONS:
Overall Officials: Wensha Yang, Ph.D., Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States